CLINICAL TRIAL: NCT01152294
Title: Measuring Quality of Decisions About Treatment of Menopausal Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Boston (Other)
Collaborators: Foundation for Informed Medical Decision Making (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Carol Cosenza, Project Manager, University of Massachusetts, Boston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CSR-DQ1-001
Record Dates: First submitted 2010-06-22; First posted 2010-06-29 (Estimated); Results first posted 2012-08-20 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-07

CONDITIONS: Menopause
Keywords: Menopause; Decision making; Decision aids; Decision quality instrument
MeSH Terms: interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Group not receiving the decision aid (DVD and booklet)
- Decision Aid (Experimental): Group receiving the decision aid (DVD/booklet)
  Interventions: Behavioral: DVD & Booklet called: Managing Menopause

INTERVENTIONS:
Behavioral: DVD & Booklet called: Managing Menopause — DVD and booklet that provides information about treatment choices for menopause symptoms. Complete title: Managing Menopause: Choosing treatments for menopause symptoms
  Other Names: Decision aids; Shared decision making programs
  Arms: Decision Aid

SUMMARY:
The purpose of this randomized controlled trial is to examine the impact of a patient decision aid on the quality of decisions about managing symptoms of menopause. In particular, we will examine whether the decision aid increases knowledge about menopause/managing menopause symptoms and concordance between goals and treatment choices.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 40-60
* Talked with health care provider about ways to manage menopause within last year OR seriously considered taking medicine or supplement to manage menopause within the last year

Exclusion Criteria:

* Prior diagnosis of breast cancer
* Surgical or medically induced menopause (ovaries removed)

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 401 (Actual)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia M Gallagher, PhD, Study Director — University of Massachusetts, Boston; Karen R Sepucha, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Center for Survey Research - University of Massachusetts Boston, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through online and newspaper ads by the Center for Survey Research in 17 cities: Atlanta, Baltimore, Boston, Chicago, Dallas-Ft. Worth, Denver, Detroit, Ft. Myers, Houston, Los Angeles, Minneapolis, New York, Phoenix, Portland, Raleigh-Durham, San Francisco, Washington, D.C.
Pre-assignment Details: Participants were randomized to receive a DVD and booklet or no DVD and to participate by phone or IVR (automated telephone survey system).
Period: Overall Study
Arm/Group | Control | Decision Aid
Started | 213 | 188
Completed | 213 | 188
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Decision Aid | Total
Number analyzed (Participants) | 213 | 188 | 401
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 212 | 186 | 398
  >=65 years | 1 | 2 | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 51 (5.1) | 51 (5.5) | 51 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 213 | 188 | 401
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 213 | 188 | 401

OUTCOME MEASURES:

1. Primary Outcome: Menopause Knowledge
Description: Total knowledge score from factual questions about menopause and methods for managing menopause symptoms. Score is the percent of knowledge questions answered correctly (0 - 100%)
Time Frame: 2 weeks, on average
Population: Participants were randomized to not receive the decision aid (DVD and booklet)or to receive the decision aid and booklet.
Measure: Mean (Standard Deviation); unit: Percentage (0-100%)
Arm/Group | Control | Decision Aid
Number analyzed (Participants) | 199 | 182
Percentage (0-100%) | 51.3 (16.0) | 55.8 (18.4)
Statistical Analysis 1: Comparison: Control vs Decision Aid; We tested for a difference in the mean total knowledge score between the decision aid and control groups using independent t-test (2 sided). With 100 patients in each arm, the study had more than 90% power to detect a 10% difference in knowledge assuming a common standard deviation of 18%; Test type: Superiority or Other; p = 0.01, t-test, 2 sided; Mean Difference (Net) = 4.6, 95% CI 2-sided [1.02 to 7.96], Standard Deviation 2.4

2. Secondary Outcome: Value Concordance
Description: Measure of how concordant respondents' actual decisions about treatment for their menopause symptoms are with their stated beliefs
Time Frame: 2 weeks, on average
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: August 10, 2010 to December 2, 2010
Arm/Group | Control | Decision Aid
Serious Adverse Events (participants affected / at risk) | 0/213 | 0/188
Other Adverse Events (participants affected / at risk) | 0/213 | 0/188

LIMITATIONS AND CAVEATS:
Participants who answered less than half the knowledge questions do not have a total knowledge score (primary outcome).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No